CLINICAL TRIAL: NCT00505856
Title: Dermabond Skin Adhesives vs Skin Staples for Closure of Repeat Cesarean Section Skin Incisions
Status: Terminated | Type: Observational
Why Stopped: Resident project--resident left institution and was not picked up by anyone else
Sponsor: Texas Tech University Health Sciences Center (Other)
Other Study IDs: L06-158
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Last update posted 2008-12-12 (Estimated); Status verified 2008-12

CONDITIONS: Pregnancy

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The use of dermabond skin adhesive vs. skin staples for the closure of repeat c-section incisions.

DETAILED DESCRIPTION:
This research is interested in using Dermabond skin adhesive as a closure for repeat cesarean incisions. The current standard of practice is to close these incisions with either skin surgical staples or suture. We will compare the use of Dermabond vs. the use of skin surgical staples in the closure of these incisions.

Eightenn-50 year old pregnant patients are eligible for this study. Other inclusion criteria are history of a previous Pfannenstiel (transverse) incision and no evidence of infection at the incision site. Exclusion criteria include a previous vertical incision and active infection at the incision site. Patients will be enrolled during their prenatal appointments and the Texas Tech OB/GYN clinic, Grand Expectations, and the Southwest OB/GYN Associates offices. They will be consented by faculty, residents, and nursing staff. This is a preliminary study of 50 patients (25 in experimental arm, i.e. Dermabond and 25 in the control group, i.e. surgical skin staples). Patients will be randomized in a 1:1 fashion by placing the terms "Dermabond" and "Staples" in a sealed envelope. The envelopes will be kept in the Family Birth Center under lock and key. The envelopes will be opened at the time of repeat c-section. A data set will be collected prior to randomization and include: gravidity, parity, age, BMI (weight and height), comorbid diseases and ethnic background.

At the time of closure, there will be subcutaneous reapproximation of tissue to take the tension off of the skin. This will occur for all subjects. The type of suture used and the suturing technique will be recorded. The skin edges will be closed with either Dermabond per label directions or with skin staples, depending on randomization. The length of the incision, the type of suture used, the type of stitch used and the total number of layers closed will also be documented. The number of staples will also be documented.

During the hospital stay, the patients wound will be examined on post operative day one and three. At this time, wound characteristics will be documented using a modified Hollander scale. A digital photograph of the incision will also be taken. The patient will also be given a patient satisfaction survey about their wound. The patients will then be seen at two weeks post partum and again at six weeks post partum. The wound characteristics and patient satisfaction will again be documented using the above materials.

Other data that will be collected includes the incidence of wound infection, as documented by wound culture, wound separation rates as documented by need for wound packing and wound dehiscence.

ELIGIBILITY:
Inclusion Criteria:

* pregant; between ages of 18-50; previous cesarean section with a transverse (sideways) skin incision.

Exclusion Criteria:

* Previous vertical (Up and Down) skin incision; active infection at site of incison

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-07; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Casanova, MD, Principal Investigator — Texas Tech University
Locations (1):
- Texas Tech University HSC Dept OB/GYN, Lubbock, Texas, United States